CLINICAL TRIAL: NCT02577549
Title: Weight Loss and Exercise for Communities With Arthritis in North Carolina
Acronym: WE-CAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00033618.WE-CAN; U01AR068658 (NIH)
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Results first posted 2023-03-15 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis
Keywords: Knee Pain; Exercise; Diet; Weight Loss
MeSH Terms: conditions — Osteoarthritis; Motor Activity; Weight Loss | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet & Exercise (Experimental): Participants will attend an exercise class 3 days/week for 18 months. The exercise program will consist of a 15-minute aerobic phase, a 20-minute strength training phase, a second 15-minute aerobic phase, and a 10 minute cool down phase. Participant's will also attend individual and group diet sessions. Each participant's minimum weight loss goal will be 10% of baseline body weight.
  Interventions: Behavioral: Diet & Exercise
- Attention Control (Active Comparator): The attention control intervention will cover an 18-month period. There will be five total face to face group meetings over the 18 months, with one meeting each at months 1, 3, 6, 9, and 15; and during the other months (months 2-5, 7-11, 13-17) participants will receive a combination of informational packets, webinars, phone sessions, and/or emails based on continued monitoring of participant needs and delivered via their preferred mode of contact.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Diet & Exercise — Participants will attend exercise and diet classes.
  Arms: Diet & Exercise
Behavioral: Attention Control — Participants will attend healthy living classes and receive health newsletters and phone calls/emails/texts.
  Arms: Attention Control

SUMMARY:
This study aims to develop and demonstrate the effectiveness of a systematic, practical, cost-effective diet-induced weight loss and exercise intervention in both urban and rural communities that can reduce pain and improve other clinical outcomes in knee OA patients. This pragmatic community-based trial will determine if the investigators previous findings translate to real-world settings and will address common concerns about barriers to effectiveness/ implementation.

DETAILED DESCRIPTION:
Obesity is a modifiable risk factor for knee osteoarthritis (OA), and weight loss is an effective non-pharmacologic treatment to reduce pain. Recently, the investigators determined that under ideal, highly controlled circumstances, a diet-induced weight loss of 10% combined with exercise was significantly better at reducing pain than either intervention alone. Compared to the investigators previous longterm weight loss and exercise trials of knee OA, the diet-induced weight loss and exercise group was twice as effective at relieving pain. Whether the investigators results can be generalized to less rigorously monitored patient cohorts is unknown. Thus the challenge the investigators now face is to provide the practical means to implement this proven treatment in the community setting. This study aims to develop and demonstrate the effectiveness of a systematic, practical, cost-effective diet-induced weight loss and exercise intervention in both urban and rural communities that can reduce pain and improve other clinical outcomes in knee OA patients. This pragmatic community-based trial will determine if the investigators previous findings translate to real-world settings and will address common concerns about barriers to effectiveness/ implementation.

Participants will be 820 ambulatory, community-dwelling, overweight and obese men and women who meet the American College of Rheumatology clinical criteria for knee OA. The primary aim is to determine whether a pragmatic, community-based 18-month diet-induced weight loss and exercise intervention implemented in three North Carolina counties with diverse residential (from urban to rural) and socioeconomic composition significantly decreases knee pain in overweight and obese adults with knee OA relative to an attention control group. Secondary aims will determine whether this intervention improves self-reported function, health-related quality of life, and mobility. The investigators will also establish the cost-effectiveness of this pragmatic, community-based, multimodal diet-induced weight-loss and exercise program by conducting cost-effectiveness and budgetary impact analyses using data from the current trial in a validated computer-simulated model of knee OA.

Many physicians who treat people with knee OA have no practical means to implement weight loss and exercise treatments. This study is significant in that it will test the effectiveness of a long-awaited and much needed community-based program that will serve as a blueprint for clinicians and public health officials in both urban and rural communities to implement a weight loss and exercise program designed to reduce knee pain and improve other clinical outcomes in overweight and obese people with knee OA that can be sustained long-term and at a reasonable cost.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 50
* Knee Pain plus American College of Rheumatology (ACR) Criteria for Knee Osteoarthritis
* BMI = 27 ≥ kg/m2

Exclusion Criteria:

* Significant co-morbid disease that would threaten safety or impair ability to participate in interventions or testing (Blindness; Type 1 diabetes; Severe coronary artery disease)
* Not sufficiently overweight or obese, BMI < 27 kg/m2
* Not having knee pain
* Inability to finish 18-month study or unlikely to be compliant (Planning to leave area > 2 month during the next 18 months; Unwilling to change eating or physical activity habits; Unwilling to discontinue pain medication use for 3 days prior to testing visit)
* Age, age < 50
* Other conditions that may prohibit the effective delivery of the intervention (Unable to provide own transportation to exercise center; Unable to read or write)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2016-01; Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Messier, PhD, Principal Investigator — Wake Forest University; Leigh Callahan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (3):
- United States (3):
  - Johnston County - UNC Chapel Hill, Chapel Hill, North Carolina
  - Haywood County - Haywood Regional Medical Center, Waynesville, North Carolina
  - Forsyth County - Wake Forest University/Wake Forest University Health Sciences, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messier SP, Callahan LF, Beavers DP, Queen K, Mihalko SL, Miller GD, Losina E, Katz JN, Loeser RF, Quandt SA, DeVita P, Hunter DJ, Lyles MF, Newman J, Hackney B, Jordan JM. Weight-loss and exercise for communities with arthritis in North Carolina (we-can): design and rationale of a pragmatic, assessor-blinded, randomized controlled trial. BMC Musculoskelet Disord. 2017 Feb 22;18(1):91. doi: 10.1186/s12891-017-1441-4. PMID 28228115
- [Result] Messier SP, Beavers DP, Queen K, Mihalko SL, Miller GD, Losina E, Katz JN, Loeser RF, DeVita P, Hunter DJ, Newman JJ, Quandt SA, Lyles MF, Jordan JM, Callahan LF. Effect of Diet and Exercise on Knee Pain in Patients With Osteoarthritis and Overweight or Obesity: A Randomized Clinical Trial. JAMA. 2022 Dec 13;328(22):2242-2251. doi: 10.1001/jama.2022.21893. PMID 36511925
- [Derived] Messier SP, Gill ME, Mihalko SL, Beavers DP, Queen K, Miller GD, Losina E, Katz JN, Loeser RF, DeVita P, Hunter DJ, Quandt SA, Lyles MF, Hudson D, Callahan LF. Clinical, Health-Related Quality of Life, and Gait Differences Among Obesity Classes in Adults With Knee Osteoarthritis. Arthritis Care Res (Hoboken). 2024 Apr;76(4):503-510. doi: 10.1002/acr.25265. Epub 2024 Jan 16. PMID 37885103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We used overlapping recruitment strategies. A combination of mailings, local newspaper ads, and direct targeting through electronic health records were used. We also had strong ties with local aging service networks and access to senior centers, senior high-rise residential sites, churches, and a large database of older adults who signed consent to be contacted about participating in future clinical trials.
Groups:
- Diet & Exercise: Participants attended an exercise class 3 days/week for 18 months. The exercise program consisted of a 15-minute aerobic phase, a 20-minute strength training phase, a second 15-minute aerobic phase, and a 10 minute cool down phase. Participant's also attended individual and group diet sessions. Each participant's minimum weight loss goal was 10% of baseline body weight.
- Attention Control: The attention control intervention covered an 18-month period delivered in five
  1-hour, in-person group meetings at months 1, 3, 6, 9, and 15. Information was also provided in paper packets and in individual telephone sessions every other month.
Period: Overall Study
Arm/Group | Diet & Exercise | Attention Control
Started | 414 | 409
Completed | 336 | 332
Not Completed | 78 | 77

BASELINE CHARACTERISTICS:
Groups:
- Diet & Exercise: Participants attended an exercise class 3 days/week for 18 months. The exercise program consisted of a 15-minute aerobic phase, a 20-minute strength training phase, a second 15-minute aerobic phase, and a 10 minute cool down phase. Participant's also attended individual and group diet sessions. Each participant's minimum weight loss goal was 10% of baseline body weight.
  Diet & Exercise: Participants attended exercise and diet classes.
- Attention Control: The attention control intervention covered an 18-month period delivered in five 1-hour, in-person group meetings at months 1, 3, 6, 9, and 15. Information was also provided in paper packets and in individual telephone sessions every other month.
  Attention Control: Participants attended healthy living classes and received health newsletters and phone calls/emails/texts.
- Total: Total of all reporting groups
Arm/Group | Diet & Exercise | Attention Control | Total
Number analyzed (Participants) | 414 | 409 | 823
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (7.8) | 64.7 (7.8) | 64.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 320 | 317 | 637
  Male | 94 | 92 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 407 | 401 | 808
  Unknown or Not Reported | 0 | 5 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 111 | 116 | 227
  White | 289 | 281 | 570
  More than one race | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Womac pain score [Mean (Standard Deviation); unit: score on a scale] — Range, 0 to 20 (0, no pain; 2 to 8, mild; >8 to 14, moderate; and >14 to 20, severe); between-group Minimal clinically important differences (MCID) = 1.6, calculated as half the Standard Deviation (SD).
  score on a scale | 7.5 (3.2) | 7.5 (3.3) | 7.5 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Knee Pain
Description: To determine whether a pragmatic, community-based, 18-month diet-induced weight-loss and exercise intervention implemented in three North Carolina counties with diverse residential (from urban to rural) and socioeconomic composition significantly decreases knee pain [as measured by the Western Ontario McMasters Universities Osteoarthritis Index (WOMAC) pain subscale] in overweight and obese adults with knee Osteoarthritis (OA) compared to an attention-control group - test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4) - Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations - The WOMAC measures five items for pain (score range 0-20). Measure Description: Range, 0 to 20 (0, no pain; 2 to 8, mild; >8 to 14, moderate; and >14 to 20, severe); between-group MCID = 1.6, calculated as half the SD.
Time Frame: 18 months
Population: A total of 13 persons (7 in D&E and 6 in attention control) did not complete this testing measure but completed other measures.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Diet & Exercise | Attention Control
Number analyzed (Participants) | 329 | 316
score on a scale | 5.0 [4.6 to 5.4] | 5.5 [5.1 to 5.9]

2. Secondary Outcome: Function
Description: To determine whether a pragmatic, community-based, 18-month, diet-induced weight-loss and exercise intervention improves WOMAC self-reported function in overweight and obese adults with knee OA compared to an attention control group - test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4) - Higher scores on the WOMAC indicate more pain, stiffness, and functional limitations. The WOMAC function score is a total of seventeen items for function (total score range 0-68). Measure Description: Range, 0 to 68 (0, no difficulty; 68, extreme).
Time Frame: 18 months
Population: Not all persons completing the study completed this measure at follow up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Diet & Exercise | Attention Control
Number analyzed (Participants) | 325 | 311
score on a scale | 16.5 [15.3 to 17.7] | 19.8 [18.6 to 21.0]

3. Secondary Outcome: Health Related Quality of Life (SF-36) Physical Subscale
Description: To determine whether a pragmatic, community-based, 18-month, diet-induced weight-loss and exercise intervention improves health-related quality of life as measured by the physical subscale of the SF-36 questionnaire in overweight and obese adults with knee OA compared to an attention control group - Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state - The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Time Frame: 18 months
Population: Not all persons completing the study completed this measure at follow up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Diet & Exercise | Attention Control
Number analyzed (Participants) | 321 | 306
score on a scale | 41.4 [40.2 to 42.6] | 37.6 [36.3 to 38.8]

4. Secondary Outcome: Mobility (Six Minute Walk)
Description: To determine whether a pragmatic, community-based, 18-month, diet-induced weight-loss and exercise intervention improves 6-minute walk distance (an accepted measure of mobility) in overweight and obese adults with knee OA compared to an attention control group.
Time Frame: 18 months
Population: Not all persons completing the study completed this measure at follow up.
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Diet & Exercise | Attention Control
Number analyzed (Participants) | 247 | 219
meters | 419 [411 to 428] | 376 [368 to 385]

5. Other Pre Specified Outcome: Cost-effectiveness
Description: To establish the cost-effectiveness of this pragmatic, community-based, multimodal diet-induced weight-loss and exercise program by conducting cost-effectiveness and budgetary impact analyses using data from the current trial in a validated computer-simulated model of knee OA.
Time Frame: 18 months
Population: Currently only data for the primary outcome and some of the secondary outcomes have been analyzed and published. Additional analyses are being conducted. The cost effectiveness outcome measure will be available to report in the coming months.
Arm/Group | Diet & Exercise | Attention Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from after the participant was randomized until completion of the 18 month intervention.
Arm/Group | Diet & Exercise | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/414 | 3/409
Serious Adverse Events (participants affected / at risk) | 67/414 | 96/409
Other Adverse Events (participants affected / at risk) | 107/414 | 93/409
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diet & Exercise (N=414) | Attention Control (N=409)
Car Accident (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Surgery Complications (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ruptured Blood Vessel (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gall Bladder Surgery (Surgical and medical procedures) | 2 (2) | 2 (2)
Bariatric Surgery (Surgical and medical procedures) | 1 (1) | 3 (3)
Hip Replacement (Surgical and medical procedures) | 1 (1) | 3 (3)
Cardiac Monitor (Surgical and medical procedures) | 2 (2) | 0 (0)
Other Knee Surgery (Surgical and medical procedures) | 2 (2) | 0 (0)
Knee replacement (Surgical and medical procedures) | 17 (19) | 23 (23)
Hernia Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Knee Amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Oophorectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Throat Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Appendectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac Ablation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Intestinal Blockage Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Neck Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Shoulder Replacement Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Numbness/Tingling (Nervous system disorders) | 1 (1) | 0 (0)
Fainting/Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1)
Mood Alteration (Psychiatric disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Low Blood Sodium (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 4 (4) | 4 (5)
Chest Pain (Cardiac disorders) | 2 (2) | 4 (4)
Stroke (Cardiac disorders) | 5 (5) | 0 (0)
Heart Attack (Cardiac disorders) | 1 (1) | 2 (3)
TIA (Cardiac disorders) | 1 (1) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 2 (2)
AV Heart Block (Cardiac disorders) | 1 (1) | 0 (0)
Blood Clot (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia & Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Cardiac disorders) | 0 (0) | 1 (1)
Bowel Obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ketoacidotic Coma (Gastrointestinal disorders) | 0 (0) | 1 (1)
UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
Colovesical Fistulitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Enlarged Prostate (Renal and urinary disorders) | 0 (0) | 1 (1)
Cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Impaired Kidney Function (Renal and urinary disorders) | 0 (0) | 1 (1)
Cancer (Blood and lymphatic system disorders) | 7 (7) | 9 (9)
Tumor (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Elevated PSA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Rapid Weight Loss (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 1 (1) | 0 (0)
Breathing Difficulty (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure and Coronary Artery Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (3)
Septic Shock (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Streptococcal Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Finger Infection (Infections and infestations) | 1 (1) | 0 (0)
Intestinal Infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diet & Exercise (N=414) | Attention Control (N=409)
Fall (Injury, poisoning and procedural complications) | 71 (85) | 37 (46)
Knee Injection (Surgical and medical procedures) | 36 (44) | 56 (75)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT02577549/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT02577549/ICF_002.pdf